CLINICAL TRIAL: NCT01216891
Title: Recovery After an Initial Schizophrenia Episode (RAISE): The RAISE Connection Program Duration of Untreated Psychosis (DUP)
Brief Title: Multi-disciplinary Treatment for Patients Experiencing First Episode of Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Maryland (Other); New York State Office of Mental Health (OMH) (Unknown); Maryland Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Lisa Dixon, Director Center for Practice Innovations, Research Foundation for Mental Hygiene, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAISE Connection; HHSN271200900020C (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Delusional Disorder; Psychosis
Keywords: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Delusional Disorder; Psychosis; First episode
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Team-based treatment (Experimental)
  Interventions: Behavioral: Multi-element, team-oriented treatment

INTERVENTIONS:
Behavioral: Multi-element, team-oriented treatment — Participants will receive treatment and services based on their needs coordinated by a small team that is led by a clinical coordinator. Services that are available to the participants include social skills training, medication treatment to address symptoms, education and employment advising, and substance use treatment.

SUMMARY:
This study will assess the effectiveness of an experimental treatment intervention for adolescents and adults who have experienced their first episode of psychosis during the past two years.

The DUP sub-study will collect pathways to care information that will be used to inform the development and pilot testing of strategies that aim to reduce DUP among individuals experiencing a first episode of psychosis.

DETAILED DESCRIPTION:
This study is part of the National Institute of Mental Health's Recovery After an Initial Schizophrenia Episode (RAISE) Project. The RAISE Project seeks to fundamentally change the trajectory and prognosis of schizophrenia through coordinated and aggressive treatment in the earliest stages of illness. This study, the RAISE Connection Program, is one of the two independent research studies that NIMH has funded to conduct the NIMH RAISE Project. The Connection Program is being supported in whole or in part with Federal funds from the American Recovery and Reinvestment Act of 2009 and the NIMH, National Institutes of Health, Department of Health and Human Services. The Connection Program aims to to assess the effectiveness of a Team-based intervention for individuals with a first psychotic episode, observing outcomes over time for our study participants. When tracking outcomes, the Connection Program will make comparisons with what is known about the natural history of untreated first episode of psychosis as well as usual care outcomes from other experimental studies.

This study is for people who have experienced symptoms such as hallucinations, unusual thoughts or beliefs, or disorganized thinking for the first time during the past two years. Without treatment, many people have a difficult time with these symptoms, which can be very upsetting and also make it hard to socialize, study, or work.

People have different wishes and needs, and it is not clear what combination of treatments and services is best for any one person. There are many possible treatments and services, such as medications, talk therapy, case management, and school and job counseling. This study will adapt and evaluate the impact of a comprehensive and integrated treatment intervention for first episode psychosis to be delivered in real-world practice settings to promote symptomatic recovery, minimize disability, and maximize social, academic, and vocational functioning.

Participation in this study will last up to 2 years. At the baseline visit, participants will be enrolled to receive the experimental intervention. During the study period, participants will take part in research interviews every three to six months for a total of 6 interviews. Each of these research interviews will take 1.5 to 3 hours to complete. Assessments of participants' health condition, overall function and illness severity, employment status, academic performance, and social functioning will be conducted during these research interviews. In addition to assessing functioning and illness severity, this study will also address substance abuse and utilization of healthcare services. Participants will also be measured for their height, weight and waist circumference. This portion of the study concluded in December 2013.

The RAISE-DUP contract modification seeks additional information on the referral pathways that resulted in enrollment in the RAISE Connection Program from individuals who participated in RAISE Connection Program services and their family members. Information gathered through qualitative research interviews will be used to inform the development and pilot testing of outreach, education, and engagement intervention strategies, to serve the larger goal of reducing the duration of untreated psychosis among individuals experiencing a first episode of psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 15-35 years old (16-35 years old in New York)
* Diagnosis of schizophrenia, schizoaffective and schizophreniform disorder, delusional disorder, or psychosis not otherwise specified (NOS)
* Duration of psychotic symptoms > 1 week and < 2 years
* Ability to provide informed consent
* Ability to speak and understand English
* Anticipated availability to participate in the intervention for at least 1 year
* RAISE-DUP: participants must have been enrolled in the RAISE study

Exclusion Criteria:

* Medical conditions which impair function independent of psychosis
* Other diagnoses associated with psychosis:
* Substance-induced psychotic disorder
* Psychotic affective disorder (major depressive or manic episode with psychotic features)
* Psychotic disorder due to a general medication condition
* Mental retardation

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The Mental Illness Research Education and Clinical Center Global Assessment of Functioning (MIRECC GAF) | Measured at baseline
  This measures occupational functioning, social functioning and symptom severity.
The Mental Illness Research Education and Clinical Center Global Assessment of Functioning (MIRECC GAF) | Measured at Month 6
The Mental Illness Research Education and Clinical Center Global Assessment of Functioning (MIRECC GAF) | Measured at Month 12
The Mental Illness Research Education and Clinical Center Global Assessment of Functioning (MIRECC GAF) | Measured at Month 18
The Mental Illness Research Education and Clinical Center Global Assessment of Functioning (MIRECC GAF) | Measured at Month 24
Pathways to Care Qualitative Interview | Measured at baseline
  This assessment gathers information on help-seeking events and participant recommendations.

SECONDARY OUTCOMES:
The Clinical Global Impression (CGI) - Severity scale | Measured at baseline
  This assesses the level of severity of illness.
Calgary Depression Scale | Measured at baseline
  This assesses depression in people with schizophrenia.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Measured at baseline
  This measures the presence and severity of symptoms of schizophrenia.
The Clinical Global Impression (CGI) - Severity scale | Measured at Month 6
  This assesses the level of severity of illness.
The Clinical Global Impression (CGI) - Severity scale | Measured at Month 12
  This assesses the level of severity of illness.
The Clinical Global Impression (CGI) - Severity scale | Measured at Month 18
  This assesses the level of severity of illness.
The Clinical Global Impression (CGI) - Severity scale | Measured at Month 24
  This assesses the level of severity of illness.
Calgary Depression Scale | Measured at Month 6
  This assesses depression in people with schizophrenia.
Calgary Depression Scale | Measured at Month 12
  This assesses depression in people with schizophrenia.
Calgary Depression Scale | Measured at Month 18
  This assesses depression in people with schizophrenia.
Calgary Depression Scale | Measured at Month 24
  This assesses depression in people with schizophrenia.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Measured at Month 6
  This measures the presence and severity of symptoms of schizophrenia.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Measured at Month 12
  This measures the presence and severity of symptoms of schizophrenia.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Measured at Month 18
  This measures the presence and severity of symptoms of schizophrenia.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Measured at Month 24
  This measures the presence and severity of symptoms of schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dixon, MD, Principal Investigator — Columbia University; Melanie Bennett, PhD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Carruthers Clinic, Baltimore, Maryland
  - Washington Heights Community Service Clinic, New York, New York

REFERENCES:
- See also: Related Info — http://www.nimh.nih.gov/RAISE